CLINICAL TRIAL: NCT03904342
Title: Comparing the Sophie RA-CBT System and Telemedically-delivered CBT: a Pilot Implementation Study
Brief Title: Sophie Pilot Implementation and Assessment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not conducted due to concerns about collaboration with an outside vendor for the control condition.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-37919; 4153360 (Other Grant/Funding Number: CIIS Evans Center)
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Depression Chronic; Advanced Cancer; Anxiety
Keywords: Cognitive behavioral therapy (CBT); Sophie CBT; iHope CBT; Consolidated Framework for Implementation Research (CFIR)
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sophie CBT (Active Comparator): The Sophie Cognitive Behavioral Therapy (CBT) intervention is a tablet-based computerized CBT and self-management education intervention that consists of an evidence-based cognitive behavioral therapy self-management curriculum divided into 6 discrete modules. Patients will have up to 8 weeks to work through the modules on the tablet.
  Interventions: Behavioral: Sophie CBT System
- iHope CBT (Active Comparator): iHope CBT is a telemedically-delivered CBT package. The iHope system comprises a HIPAA-compliant platform on which real, live, licensed clinicians provide cognitive behavioral therapy via video conferencing, phone calls, and text messaging. iHope will be delivered on subjects' preferred electronic device (mobile phone, laptop, tablet).
  Interventions: Behavioral: iHope CBT

INTERVENTIONS:
Behavioral: Sophie CBT System — The Sophie CBT system is a tablet-based system that delivers self-paced cognitive behavioral therapy educational curriculum in the format of 6 discrete modules.
  Arms: Sophie CBT
Behavioral: iHope CBT — Licensed therapists will use the iHope HIPAA-compliant telemedicine platform to deliver cognitive behavioral therapy to patients via telephone, videoconferencing, and/or text chat.
  Arms: iHope CBT

SUMMARY:
Evidence-based interventions using cognitive behavioral therapy (CBT) and self-management education have been demonstrated to effectively treat symptoms of depression and improve the quality of life in populations with chronic illness. Research indicates that CBT is the most effective psychosocial treatment for depression; as effective as pharmacotherapy and as effective as adding another medication for patients who do not respond to one antidepressant alone. Despite the existence of proven efficacious treatments for depression, however, fewer than half of patients for whom depression treatment is indicated receive the services they need. Access barriers (i.e., transportation, insurance coverage), limited clinician availability (i.e., long waitlists, difficulty finding a provider), and competing (and time-consuming) medical priorities contribute to inadequate depression treatment for individuals with serious chronic illness. In this research the investigators will conduct a pilot randomized trial to compare results from implementation of two CBT strategies iHope and Sophie.

DETAILED DESCRIPTION:
A pre-implementation pilot study will be conducted with 20 adult patients diagnosed with advanced (Stage 3 or 4) cancer who screen positive for moderate depression and are receiving care at the Solomont Center for Hematology and Medical Oncology at Boston Medical Center (BMC) with the following specific aims:

1. Using the Consolidated Framework for Implementation Research (CFIR) as a guide, design a pilot implementation strategy for introducing the Sophie CBT system and iHope system into the clinical context of care (Months 1-4)
2. Conduct a pre-implementation pilot study with randomization of 20 cancer patients who screen positive for depression and/or anxiety into two arms with Sophie CBT or iHope telemedicine (10 participants each) to: a) assess the feasibility, acceptability, and appropriateness of implementing the Sophie CBT and iHope interventions in an ambulatory cancer treatment center and b) evaluate the potential impact of the Sophie CBT and iHope interventions on measures of depression, anxiety, coping, and quality of life for cancer patients with comorbid depression (Months 5-10)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage 3 or 4 cancer receiving care at Solomont Cancer Center
* GAD score >10 AND/OR positive screening for moderate to severe depressive symptoms (PHQ-8>9).
* Comfortable using tablet, phone and computer
* Has telephone access
* Speaks English
* Lives in greater Boston area

Exclusion Criteria:

* Patients without the capacity to provide informed consent
* Ongoing substance use disorder
* Patients with Schizophrenia and Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | baseline, 8 weeks
  Changes in depressive symptoms will be measured using the PHQ-8, which is an 8-item scale with scores ranging from 0 to 24, with higher scores indicative of more depressive symptoms

SECONDARY OUTCOMES:
Change in anxiety | baseline, 8 weeks
  The Generalized Anxiety Disorder 7 (GAD-7) will be used to assess changes in anxiety. The GAD-7 is a 7-item questionnaire that asks how often an individual has been bothered by a given item over the last 2 weeks. Scores range from 0 ("not at all") to 3 ("nearly every day.") A higher overall score indicates a greater level of anxiety.
Change in coping | baseline, 8 weeks
  Changes in coping will be assessed using the Ways of Coping scale which is a 66 item scale with potential responses from 1 to 4, with higher scores indicative of more frequent use of a particular strategy.
Changes in quality of life | baseline, 8 weeks
  Changes in quality of life will be assessed using the Quality of Life Scale (QOLS), which is a 15-item scale with potential responses ranging from 1 to 7, with higher scores indicating a higher level of satisfaction with quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Mitchell, MD, Principal Investigator — Boston Medical Center

IPD SHARING:
Plan to Share IPD: No